CLINICAL TRIAL: NCT03809741
Title: Prevention of Neonatal and Maternal Infection During Labor and Delivery in Rural Healthcare Sites in Zambia - Intervention Phase
Brief Title: Intervention Zambia Rural L&D Infection Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: Right to Care (Other); Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: H-38261
Record Dates: First submitted 2019-01-14; First posted 2019-01-18 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Postpartum Infection; Neonatal Infection
Keywords: Infection prevention and control; Alcoholic hand rubs; Intrapartum care; Postpartum care; Infection Control Assessment Tool (ICAT); Rural Zambia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Preventing L&D Infections (Experimental): Low-cost bundled L&D infection prevention interventions will be implemented, including education, visual reminders, feedback, and alcoholic hand rub supply. Infection control practices and child delivery outcomes will be assessed after implementation of these interventions.
  Interventions: Other: Bundled L&D Infection Prevention Interventions

INTERVENTIONS:
Other: Bundled L&D Infection Prevention Interventions — The following bundle of infection prevention interventions will be implemented at each study site for 12 weeks:
  Education: 2 day module of Infection Prevention and Control (IPC) training and education at the beginning of the period, with specific information pertaining to labor and delivery. A refresher course will be administered at week 6.
  Feedback: Monthly feedback sessions detailing IPC practices
  Reminders: Visual poster reminders on hand hygiene and daily SMS reminders on best practices for peripartum and postnatal care.
  Alcohol Hand Rub (AHR) supply: Provision of AHR, produced by WHO standards and guides in collaboration with district pharmacy

SUMMARY:
This is the intervention phase of a study to investigate the impact of low-cost bundled interventions on improving the infection control practices in the labor and delivery units in rural healthcare settings in Zambia. A baseline observational phase of the health care providers' infection control procedures was done. In this intervention phase, low-cost bundle of interventions, including health care provider education, behavior feedback, visual and Short Message Service (SMS)/text message reminders, and provision of alcoholic hand rubs, will be implemented at 5 study sites. 12 weeks after the initiation of interventions, endline data will be collected. The data from endline after interventions will be compared with baseline data from observational phase to detect changes in infection control practices at each study site after the interventions.

DETAILED DESCRIPTION:
The total duration of the intervention phase is estimated to be 4 months. During this time, the investigators will collaborate with the healthcare workers (HCWs) at each study site and the district pharmacist.

The study team will visit each site separately and administer the training modules on-site during the first month of the research until all of the modules have been completed for all of the Labor and Delivery (L&D) staff, which usually consist of about 2-3 people. A quiz will be administered before and after the training session to assess change in knowledge after the training.

SMS reminders will be sent every weekday to promote best infection control practices in the L&D. Posters will also be posted for visual reminders of best practices around the health center.

After the initial training, each health centers will be visited twice a month by a study team member to assess alcohol rubs (AHR) stock, gather feedback and comments, and evaluate postpartum maternal and neonatal infectious complications and hospital outcomes. Infection and outcome data will be shared with each site monthly. About 2 months after initial training, a refresher education and training course will be held at each study site. A quiz will be administered before and after the refresher course to assess knowledge.

The investigators will collaborate with the district pharmacy for production and distribution of AHR. The pharmacists will receive training on how to combine and mix the hand rub components per WHO guidelines, and test batches will be made prior to distribution to study sites to ensure familiarity of the pharmacy staff with its production. Quality control with an alcoholmeter will be performed with the alcohol ingredient and with the finished product, as per World Health Organization (WHO) recommendation. Afterwards, the head pharmacist will be consulted biweekly by study team member to document AHR production, budget, distribution, and any other issues.

Endline data collection will occur 12 weeks after initiation of intervention implementation. During data collection period, a study team member will meet with a L&D floor administrator in a private setting at a time convenient to the administrator to go through the questionnaire portion of the ICAT together.

Eligible pregnant women will primarily be recruited and consented outside the facility in the waiting area where they congregate prior to admission for delivery. Women who are consented will be given a "consent card" in addition to a copy of the consent form. This card will state that they have previously consented to the study, and can then be presented once they are admitted for delivery. A member of the research team will accompany the primary care provider during their provision of care and patient contact during first, second, and third stages of labor to observe, assess and document infection control behaviors and practices by the providers, using the ICAT.

A retrospective review of the logbook will be done to assess for rates of postpartum maternal and neonatal infectious complication and outcomes for participants.

During the endline data collection, an anonymous, self-administered survey will be administered to the study site HCWs to assess the knowledge, attitudes and practices of the study site HCWs towards the implemented study interventions.

ELIGIBILITY:
Inclusion Criteria for observation:

* Women of age > 15 in early first stage of labor (cervical dilation ≤ 6cm) at the study sites during the study period
* If woman is 15 to 17 must have a guardian present
* Planned vaginal delivery
* Any healthcare workers providing direct patient care to women delivering at the study sites during study period

Exclusion Criteria for observation:

* Any eligible woman who presents past the early first stage of labor (cervical dilation > 6cm)
* Woman under 18 years old without a guardian present

Inclusion criteria for logbook review:

* Women who delivered their baby at the study sites during the study period
* Newborns who were born at the study sites during the study period

Min Age: 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 37 (Actual)
Dates: Start 2019-04-11 (Actual); Primary Completion 2019-08-16 (Actual); Study Completion 2019-09-16 (Actual)

PRIMARY OUTCOMES:
Infection control practices assessed by Infection Control Assessment Tool (ICAT) score | 12 weeks
  A survey including 98 questions detailing infection control practices in the L&D. It includes questions on facility, Infection Prevention and Control (IPC) program, general IPC, hand hygiene, L&D practices, and postpartum care practices. The scores from each question on the survey will be summed for the ICAT score for each health center. Maximum score is 140 points and minimum score is 0 points, with higher score indicating better infection control practices. Of the 98 questions, 34 questions are duplicated in an observation tool in order to corroborate the accuracy of survey information by direct observation. The observation tool includes topics on supplies in the L&D and healthcare worker behaviors during childbirth. ICAT was developed by the Rational Pharmaceutical Management plus Infection Control Project team in 2009.

SECONDARY OUTCOMES:
Number of mothers with postpartum maternal infection from medical records | 12 weeks
  A mother will be counted as having postpartum maternal infection if women they have one or more of the following:sepsis, endometritis (puerperal infection), mastitis, urinary tract infection (UTI), cellulitis, and other unspecified infections documented in the medical records (ie logbook review of maternal admission, delivery, and postnatal registries).
Number of newborns with postpartum neonatal infection from medical records | 12 weeks
  A newborn will be counted as having postpartum neonatal infection if they have one or more of the following:sepsis, pneumonia, meningitis, UTI, omphalitis, and others unspecified infections documented in the medical records (ie logbook review of maternal admission, delivery, and postnatal registries).
Rates of maternal hospital outcome categories from medical records | 12 weeks
  Categories for maternal hospital outcomes include: 1) full recovery, 2) delayed discharge, 3)transfer, 4) death, and 5) no information. Information collected from logbook review of maternal admission, delivery, and postnatal registries will be assessed and the counts in each category will be divided by the total number of mothers.
Rates of neonatal hospital outcomes from medical records | 12 weeks
  Categories for neonatal hospital outcomes include: 1) full recovery, 2) delayed discharge, 3)transfer, 4) death, and 5) no information. Information collected from logbook review of maternal admission, delivery, and postnatal registries will be assessed and the counts in each category will be divided by the total number of newborns.
HCW attitudes towards infection control interventions from an anonymous survey | 12 weeks
  Summed scores from an anonymous survey designed by the investigators will be used to assess HCW (healthcare workers') attitudes towards each aspects of the interventions and the program as a whole. The survey has 28 Likert scale questions (responses range from 1 to 5 and the summed score from 28 to 140). Higher scores indicate more positive HCW attitudes toward the interventions.The survey also includes a section for any open-ended comments for each of the interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Davison Hamer, MD, Study Director — Boston University School of Public Health, Center for Global Health
Locations (5):
- Zambia (5):
  - Mangunza Rural Health Facility, Choma, Southern Province
  - Masuku Mission Rural Health Facility, Choma, Southern Province
  - Mbabala Rural Health Facility, Choma, Southern Province
  - Mochipapa Rural Health Facility, Choma, Southern Province
  - Simakutu Rural Health Facility, Choma, Southern Province

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2019-02-20): https://cdn.clinicaltrials.gov/large-docs/41/NCT03809741/ICF_000.pdf